CLINICAL TRIAL: NCT04074837
Title: Phase1a, Randomized Placebo-controlled, Single and Multiple Dose, Dose-escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Oral NNI-362 in Healthy Aged Volunteers 50 to 72 Years of Age
Brief Title: Phase1a, Dose-escalation Study of NNI-362 in Healthy Aged Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuronascent, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NNI-001; 1R01AG056561-01A1 (NIH)
Record Dates: First submitted 2019-08-27; First posted 2019-08-30 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2020-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Placebo versus NNI-362 at 10 mg, 20 mg, 60 and 120 mg liquid suspension
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcome Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo liquid suspension.
  Interventions: Drug: Placebo
- NNI-362, 10 mg (Active Comparator): NNI-362 at 10 mg in liquid suspension
  Interventions: Drug: NNI-362
- NNI-362, 20 mg (Active Comparator): NNI-362 at 20 mg in liquid suspension
  Interventions: Drug: NNI-362
- NNI-362, 60 mg (Active Comparator): NNI-362 at 60 mg in liquid suspension
  Interventions: Drug: NNI-362
- NNI-362, 120 mg (Active Comparator): NNI-362 at 120 mg in liquid suspension
  Interventions: Drug: NNI-362
- NNI-362, 240 mg (Active Comparator): NNI-362 at 240 mg in liquid suspension
  Interventions: Drug: NNI-362

INTERVENTIONS:
Drug: NNI-362 — NNI-362 small molecule in liquid suspension.
  Arms: NNI-362, 10 mg; NNI-362, 120 mg; NNI-362, 20 mg; NNI-362, 240 mg; NNI-362, 60 mg
Drug: Placebo — Placebo liquid suspension
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety, tolerability and pharmacokinetics of single and multiple doses of NNI-362 in healthy aged population.

DETAILED DESCRIPTION:
The early clinical development strategy consists of the initial evaluation of safety and tolerability of NNI-362. This FIH Phase I includes single and multiple ascending dose studies in healthy aged volunteers. Assessment of suicidal ideation/behavior will be performed at baseline and at all study visits and on days of inpatient confinement in conformance with FDA recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy aged volunteers of either sex between the ages of 50 and 72 inclusive at time of screening.

  * Subjects must be in reasonably good health as determined by investigator based on medical history, vital signs measurements, physical examination, screening laboratory results and ECG.
  * Normal age-related findings as well as well-controlled, chronic and stable medical conditions (e.g., hypertension, osteoarthritis, non-insulin dependent diabetes mellitus, osteoporosis, gout, Paget's disease, hypothyroidism) will not be exclusionary if they are not expected to compromise subject safety, study conduct, or study objectives.
  * Non-interacting medications for stable allowable medical conditions will be allowed following review and approval by the medical monitor.
  * An adequate understanding of the requirements of the study, provision of written informed consent, and agreement to abide by the study restrictions.
  * Negative urine screen for drugs of abuse within 24 h before the administration of the first dose of study drug and in the multiple dose study upon readmission to the clinical unit from outpatient status.
  * Body Mass Index (BMI) of between 18 and 30 kg/m2 inclusive, and a total body weight greater than 48kg at screening.

Exclusion Criteria:

* • Women of child-bearing potential, defined as premenopausal (unless the potential research subject has previously undergone hysterectomy and/or bilateral salpingo-oophorectomy)

  * Pregnant or breastfeeding
  * Any clinically significant hematology, chemistry, coagulation, or urinalysis value at screening and day -1 Abnormal liver enzymes (ALT and/or AST >1.5X ULN) at screening and day -1
  * Serum creatinine > ULN at screening and day -1
  * Hemoglobin <13 g/dL for males or <11.5 g/dL for females, leukocytes <3.0 X 103/uL, absolute neutrophil count <1000/uL, or platelets <150 X 103/uL at screening and day -1
  * Any significant medical illness that could compromise the interpretability of study data or affect subject safety including, but not necessarily limited to:

    * Chronic pulmonary disease or sleep apnea
    * Clinically significant cardiac arrhythmia (either at screening or based on history)
    * Congestive heart failure, valvular heart disease or ischemic heart disease
    * Pulmonary hypertension
    * Any disorder of the kidney or urinary tract
    * Active peptic ulcer disease, gastrointestinal bleeding, inflammatory bowel disease, chronic pancreatitis
    * Liver disease (excluding Gilbert's syndrome)
    * Any neurologic disorder other than chronic Bell's Palsy
    * History of malignancy that has not been cured or in complete remission for at least 10 years (excluding resected non-metastatic basal cell carcinoma)
    * History of seizure activity other than early childhood
    * Any traumatic brain injury in adulthood
  * Current smoker or nicotine user (quit less than 2 months)
  * Active substance abuse.
  * Glomerular filtration rate <50 mL/min based on Cockcroft-Gault calculation using ideal (lean) body weight or present weight.
  * Difficulty swallowing

Ages: 50 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Measure number of treatment related adverse events following single and multiple dosing of NNI-362. | 5 to 15 days
  To examine the number of participants with treatment-related adverse events according to criteria of CTCAE v4.0

SECONDARY OUTCOMES:
Measure Maximum Plasma Concentration with single or multiple dosing of NNI-362. | 48 hours
  Following single and multiple dosing of oral NNI-362 assess the maximum plasma concentration [Cmax].
Measure Area Under the Curve with single and multiple dosing of NNI-362 | 48 hours
  Following single and multiple dosing of oral NNI-362 assess the area under the curve [AUC].

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel, International, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No
This clinical trial will be available for peer-reviewed publication.

REFERENCES:
- [Derived] Kelleher-Andersson J, Yoon E, Green C, McFarlane C, Bagheri D, Thomas LP, Turner RS. First-in-human study of neuron regenerative therapy NNI-362 to evaluate the safety, pharmacokinetics, and pharmacodynamics in healthy aged population. Alzheimers Res Ther. 2025 Aug 7;17(1):185. doi: 10.1186/s13195-025-01837-0. PMID 40775373
- [Derived] Sumien N, Wells MS, Sidhu A, Wong JM, Forster MJ, Zheng QX, Kelleher-Andersson JA. Novel pharmacotherapy: NNI-362, an allosteric p70S6 kinase stimulator, reverses cognitive and neural regenerative deficits in models of aging and disease. Stem Cell Res Ther. 2021 Jan 13;12(1):59. doi: 10.1186/s13287-020-02126-3. PMID 33436007